CLINICAL TRIAL: NCT05215093
Title: Direct Access to Physiotherapy for Acute Low Back Pain: a Pragmatic Pilot Trial
Brief Title: The Direct-Physio Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: KU Leuven (Other); Universiteit Antwerpen (Other); Université Catholique de Louvain (Other); Axxon - the Belgian physiotherapy professional association (Unknown); Riziv-Inami - National Institute for the Sickness and Invalidity Insurance (Unknown)
Responsible Party: Principal Investigator, Lotte Janssens, Professor, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CME2021/066
Record Dates: First submitted 2021-12-13; First posted 2022-01-31 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Low Back Pain; Physiotherapy
Keywords: Direct access
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct physiotherapy pathway (Experimental): People with acute low back pain will directly go to a physiotherapist, who will treat the patient without prescription of the general practitioner.
  Interventions: Other: Direct access physiotherapy for acute low back pain
- Usual care pathway (Active Comparator): People with low back pain will receive usual care by the general practitioner (with or without referral to physiotherapy).
  Interventions: Other: Usual care for acute low back pain

INTERVENTIONS:
Other: Direct access physiotherapy for acute low back pain — Interventions include physiotherapeutic treatment, without prescription of the general practitioner, for low back pain according to current biopsychosocial national (KCE - Belgium) and international (NICE) guidelines.
  Arms: Direct physiotherapy pathway
Other: Usual care for acute low back pain — Interventions include standard of care by the general practitioner for low back pain according to current biopsychosocial national (KCE - Belgium) and international (NICE) guidelines.
  Arms: Usual care pathway

SUMMARY:
Previous research showed that direct access to physiotherapy, and the associated early physiotherapeutic treatment of patients with low back pain (LBP), results in improved clinical outcomes, as well as reduced health-related costs. However, despite these results, the effectiveness of direct access to physiotherapy and its impact on costs has never been investigated in Belgium. Therefore, the goal of this study is to compare the (cost-)effectiveness of direct access to physiotherapy compared to usual care by the general practitioner (GP) for patients with acute LBP.

In this study, 600 patients with acute LBP (lasting >24 hours and <6 weeks) will be divided into two groups (Dutch-speaking: n=2x150; French-speaking n= 2x150). One group will receive treatment through direct access to the physiotherapist, without prescription by a GP. The other group will follow the traditional care pathway through the GP. Th effects on pain, disability and cost-effectiveness will be analysed using questionnaires obtained before and at the end of treatment, after 3 months, after one and after two years. Primary outcomes include pain and disability. Secondary outcomes include clinical outcomes, beliefs related to LBP, quality of life, patient satisfaction, but also direct health care costs, health care resource use, as well as absenteeism and productivity loss.

The results of this study will answer the question whether direct access to physiotherapy is (cost)effective for acute LBP. In the long term, these results might be used to optimize the care pathway in Belgium for patients with acute low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-specific acute LBP defined as (based on Nicol et al. 2020):

  * pain between the 12th rib and buttocks
  * associated or not with non-dominant leg pain
* looking for LBP care for the first time in case of first episode, OR for the first time for the current episode in case of recurrent or persistent LBP
* lasting > 24 hours and < 6 weeks
* with an average pain intensity during the past 24 hours of ≥ 3 on an 11-point Numerical Pain Rating Scale
* with an Oswestry Disability Index score (version 2.1a) of at least 20% (Denteneer et al. 2018).
* Patients aged between 18 and 65 years

Exclusion Criteria:

* Recent lumbar surgery (< 1 year)
* Pregnancy
* History of (any) treatment for the current pain episode
* Red flags suggesting specific LBP (e.g. resulting from infection or neoplasm, cauda equina), based on the Belgian Health Care Knowledge Center (KCE, BEL) who published evidence-based guidelines to manage LBP and radicular pain (Van Wambeke et al. 2017), leads to exclusion from treatment within the study.
* Generalized musculoskeletal pain (based on fibromyalgia criteria) (Galvez-Sánchez and Reyes del Paso 2020).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in pain intensity | Immediately before, during the first 6 weeks and immediately after intervention and at 3 months, 1 and 2 years after enrollment
  Numeric Rating Scale
Changes in pain location and extent | Immediately before, during the first 6 weeks and immediately after intervention and at 3 months, 1 and 2 years after enrollment
  Pain Diagram of Margolis
Changes in disability | Immediately before, during the first 6 weeks and immediately after intervention and at 3 months, 1 and 2 years after enrollment
  Oswestry Disability Index

SECONDARY OUTCOMES:
Cost-effectiveness of the provided treatment (direct physiotherapy access vs usual care for acute low back pain) | Up to 2 years after enrollment
  Costs of low back pain and its treatment in terms of medical and societal costs
Changes in beliefs and cognitions related to low back | Immediately before, during the first 6 weeks and immediately after intervention and at 3 months, 1 and 2 years after enrollment
  Back Pain Attitude Questionnaire (Back-PAQ)
Changes in patient satisfaction | Immediately before, during the first 6 weeks and immediately after intervention and at 3 months, 1 and 2 years after enrollment
Changes in quality of life | Immediately before, during the first 6 weeks and immediately after intervention and at 3 months, 1 and 2 years after enrollment
  EQ-5D
Amount of / coping with flare-ups during follow-up | Immediately before, during the first 6 weeks and immediately after intervention and at 3 months, 1 and 2 years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Janssens, PhD, Principal Investigator — UHasselt
Locations (1):
- REVAL Faculty of Rehabilitation Sciences, Diepenbeek, Belgium

IPD SHARING:
Plan to Share IPD: Undecided